CLINICAL TRIAL: NCT02827617
Title: Prospective, Observational, Multi-centred, Non-interventional Study on the Identification of Biomarkers That Are Predictive of Early Ibrutinib Treatment Failure in High Risk TP53 Mutated Chronic Lymphocytic Leukemia
Brief Title: Identification of Biomarkers That Are Predictive of Early Ibrutinib Treatment Failure in High Risk TP53 Mutated Chronic Lymphocytic Leukemia
Status: Completed | Type: Observational
Sponsor: Oncology Institute of Southern Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: IOSI-EMA-001
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Ibrutinib; TP53; Chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor periphral blood cells, Plasma, Tumor genomic DNA, Plasma cell free DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TP53 mutated CLL
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Treatment with ibrutinib 420 mg quaque die in the clinical practice
  Other Names: PCI-32765

SUMMARY:
The general aim of the project is the identification of dynamic molecular markers that can help the early and real time prediction of sustained benefit or no benefit from ibrutinib treatment in CLL harboring TP53 mutations. Specific aims of the project include: 1) Assess whether clearance of TP53 mutated clones translates into a predictive biomarker of long term benefit from ibrutinib treatment in CLL. 2) Assess whether plasma cell free DNA represents a sensitive tool that can early and dynamically inform on the development of ibrutinib resistant mutations in CLL.

DETAILED DESCRIPTION:
In the chemoimmunotherapy era, TP53 mutations defined a subgroup of high risk chronic lymphocytic leukemia (CLL) patients in whom allogeneic stem cell transplantation had to be strongly considered. As a result of the accumulating favorable outcome data reported for new biological drugs, including ibrutinib, in high risk CLL harboring TP53 mutations, there is concern about whether these patients should continue to be offered allogeneic stem cell transplantation. Despite their improved outcome, a proportion of high risk CLL harboring TP53 mutations is going to develop ibrutinib resistance, which in turns translate in a very poor survival. On these bases, in the setting of ibrutinib treatment, novel biomarkers are required to re-define high risk CLL patients candidate for consolidation strategies including allogeneic stem cell transplantation. Our working hypotheses are that: i) clearance of high risk TP53 mutated clones upon treatment with ibrutinib may associate with long progression free survival (PFS), while conversely, the persistence or increase of high risk TP53 mutated subclones under ibrutinib may associate with acquisition of resistance and disease progression; and ii) plasma cell free DNA represents an accessible source of tumor DNA for the early and sensitive identification of mutations causing resistance to ibrutinib. By using highly sensitive ultra-deep next generation sequencing strategies to monitor molecular biomarkers potentially relevant for ibrutinib in DNA coming from both cellular and the plasma fractions of peripheral blood, the project has the chance of identifying new dynamic molecular markers that can help the early and real time prediction of sustained benefit from ibrutinib treatment vs imminent progression in TP53 mutated CLL patients. In the end, the results of this study will provide the bases to refine the current approach for treatment tailoring in TP53 mutated patients by allowing the identification of cases who, though being in clinical response under ibrutinib, will conceivably benefit from immediate switch to alternative options (i.e. novel drugs, allogeneic stem cell transplantation, or CART).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults 18 years or older
* Documented diagnosis of CLL, according to iwCLL 2008 criteria
* Presence of TP53 mutation as demonstrated by sequencing at the local laboratory and/or presence of 17p deletion as demonstrated by fluorescence in situ hybridization (FISH) testing performed at the local laboratory
* CLL that warrants treatment
* Planned treatment with ibrutinib 420 mg quaque die
* Willing and able to comply with scheduled visits, laboratory tests, and study procedures
* Evidence of a signed informed consent

Exclusion Criteria:

* Current or prior histological transformation from CLL to an aggressive lymphoma (ie, Richter transformation).
* Prior treatment with ibrutinib or idelalisib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult CLL patients harboring TP53 genetic abnormalities, independent of whether treatment naïve or previously treated, who warrants treatment according to iwCLL 2008 criteria, and who is planned to receive ibrutinib at standard dose as per clinical practice
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Impact of clonal response on PFS | 2/2016-2/2021
  To evaluate the impact of clonal response (namely clearance of TP53 mutated alleles in the peripheral blood (PB) CLL cells at Week 24 after treatment start) on PFS measured according to iwCLL guidelines (Hallek 2008) as the interval from ibrutinib treatment start to progression (event), death (event) or last follow-up (censoring). Progression will be defined as per investigator assessment.

SECONDARY OUTCOMES:
Proportion of clonal response at Week 24 after treatment start | 2/2016-2/2021
  To evaluate the proportion of clonal response, defined as clearance (100% reduction compared to baseline) of TP53 mutated alleles in the PB CLL cells at Week 24 after treatment start
Cumulative proportion of clonal response | 2/2016-2/2021
  To evaluate the cumulative proportion of clonal response, defined as clearance (100% reduction compared to baseline) of TP53 mutated alleles in the PB CLL cells at any time from treatment start
Impact of clonal response on overall survival | 2/2016-2/2021
  To evaluate the impact of clonal response on overall survival (OS) measured according to iwCLL guidelines (Hallek 2008) as the interval from ibrutinib treatment start to death (event) or last follow-up (censoring)
Effect of clonal response on the cumulative incidence of acquisition of resistance-mutations | 2/2016-2/2021
  To evaluate the effect of clonal response on the cumulative incidence of acquisition of resistance-mutations
Effect clonal response on the cumulative incidence of transformation to Richter syndrome | 2/2016-2/2021
  To evaluate the effect of clonal response on the cumulative incidence of transformation to Richter syndrome defined as the interval between ibrutinib treatment start to histologically documented development of an aggressive lymphoma
Impact of treatment-emergent BTK and PLCγ2 resistance mutations on PFS | 2/2016-2/2021
  To evaluate the impact of treatment-emergent BTK and PLCγ2 resistance mutations on PFS
Impact of treatment-emergent BTK and PLCγ2 resistance mutations on OS | 2/2016-2/2021
  To evaluate the impact of treatment-emergent BTK and PLCγ2 resistance mutations on OS
Impact of treatment-emergent BTK and PLCγ2 resistance mutations on the cumulative incidence of transformation to Richter syndrome | 2/2016-2/2021
  To evaluate the impact of treatment-emergent BTK and PLCγ2 resistance mutations on the cumulative incidence of transformation to Richter syndrome
Accuracy of plasma cell free DNA for the identification of BTK and PLCγ2 resistance mutations | 2/2016-2/2021
  To evaluate the sensitivity, specificity, positive predictive value, negative predictive value and accuracy of plasma cell free DNA vs tumor genomic DNA genotyping for the identification of BTK and PLCγ2 resistance mutations

CONTACTS AND LOCATIONS:
Overall Officials: Davide Rossi, MD, PhD, Principal Investigator — Oncology Institute of Southern Switzerland
Locations (13):
- Italy (9):
  - Onco Ematologia Clinico Sperimentale, I.R.C.C.S. Centro di Riferimento Oncologico, Aviano
  - Ospedale San Raffaele, Milan
  - Dipartimento di Ematologia, Niguarda Cancer Center, Ospedale Niguarda, Milan
  - Department of Medical and Surgical Sciences, section of Hematology, Modena
  - Divisione di Ematologia, Universita' del Piemonte Orientale, Novara
  - Institute of Hematology, Catholic University S. Cuore, Roma
  - Department of Haematology, Tor Vergata Hospital, Rome
  - Clinica Ematologica, Centro Trapianti e Terapie Cellulari "Carlo Melzi", Udine
  - Ematologia, Ospedale di Circolo e Fondazione Macchi, Varese
- Switzerland (4):
  - Oncology Institute of Southern Switzerland, Bellinzona, Switzerland
  - Division of Hematology, Department of Internal Medicine, Basel University Hospital, Basel
  - Hematology, Luzern Kantonsspital, Lucerne
  - Clinica Luganese Moncucco, Lugano